CLINICAL TRIAL: NCT07157046
Title: Association of q Angle and Bunion Deformity of High Heel Wearing Females of Office Working in Lahore
Status: Completed | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: DPT/Batch-Fall20/1019
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Bunion (Diagnosis)
MeSH Terms: conditions — Bunion; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Q angle was measured in association with wearing high heels in working women in offices located in Lahore. The measurement tool was Manchester scale and goniometer with a sample size of 80 people.

ELIGIBILITY:
Inclusion Criteria:

* 18-36 age
* Female
* Single leg affected
* High heel wearing

Exclusion Criteria:

* Any neurological condition
* Any laxity
* Leg length discrepancy
* Previous fracture

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Q angle was measured in association with wearing high heels in working women in offices located in Lahore
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Manchester scale | 6 Month
  It refers to two different medical assessment tools: the Manchester Scale for Hallux Valgus, which grades foot deformity severity using photographs from no deformity (Grade 1) to severe deformity (Grade 4)

CONTACTS AND LOCATIONS:
Locations (1):
- Offices in Johar Town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No